CLINICAL TRIAL: NCT01786382
Title: A Phase 1, Open-Label Study to Evaluate the Potential Effects of PPI-668 on the Pharmacokinetics of Midazolam and Omeprazole, and Potentially Telaprevir, in Healthy Adult Subjects
Brief Title: A Drug Interaction Study of the Effects of PPI-668 on the Pharmacokinetics of Midazolam and Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presidio Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PPI-668-102
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Pharmacokinetic Assessments in Healthy Volunteers
MeSH Terms: interventions — ravidasvir; Midazolam; Omeprazole; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- midazolam (Experimental): potential effects of PPI-668 on midazolam pharmacokinetics
  Interventions: Drug: PPI-668; Drug: Midazolam
- omeprazole (Experimental): potential effects of PPI-668 on omeprazole pharmacokinetics
  Interventions: Drug: PPI-668; Drug: Omeprazole
- telaprevir (Experimental): potential effects of PPI-668 on telaprevir pharmacokinetics
  Interventions: Drug: PPI-668; Drug: Telaprevir

INTERVENTIONS:
Drug: PPI-668
Drug: Midazolam
  Arms: midazolam
Drug: Omeprazole
  Arms: omeprazole
Drug: Telaprevir
  Arms: telaprevir

SUMMARY:
The primary objectives of the study are to:

* Evaluate the potential effects of PPI-668 at steady state on the pharmacokinetic (PK) profile of midazolam following a single oral dose in human subjects.
* Evaluate the potential effects of PPI-668 at steady state on the PK profile of omeprazole following a single oral dose in human subject

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legally authorized representative signs an Institutional Review Board (IRB)-approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization for sites in the United States) before any study-related procedures (including withdrawal of prohibited medication, if applicable) are performed
2. Age 18 to 50 years
3. Body mass index (BMI) 18-32 kg/m2
4. Clinical and laboratory findings consistent with good health in the opinion of the investigator
5. Women of non-childbearing potential or men who agree to utilize adequate contraception throughout the study

   1. Women of non-childbearing potential must be one of the following:

      * Postmenopausal (>2 years amenorrhea and postmenopausal status confirmed by follicle-stimulating hormone levels)
      * Surgically sterile (documentation of prior tubal ligation, hysterectomy, or oophorectomy is required)
   2. Male subjects who are not surgically sterile must agree to use one of the following birth control methods if sexually active:

      * Double-barrier contraceptive (e.g., condom plus diaphragm, condom or diaphragm with spermicidal gel/foam)
      * Female partner is at least two years postmenopausal or surgically sterile

Exclusion Criteria:

1. Positive results on any of the following tests at Screening or Day -1:

   urine pregnancy (women only), urine drugs of abuse and alcohol, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody
2. Concurrent clinically significant medical diagnosis that would potentially interfere with the subject's study compliance or confound the study results
3. Concurrent social conditions (e.g., drug or alcohol abuse, transportation difficulties) that would potentially interfere with the subject's study compliance
4. Clinically significant illness within 30 days preceding entry into the study
5. Participation in an investigational drug study within 30 days or 5 half-lives, whichever is longer, before Screening
6. Use of prescription medications within 14 days before Day 1 and throughout the study. (The use of non-prescription or over-the-counter medications is prohibited within 7 days before Day 1 and throughout the study. This includes all herbal supplements or remedies and vitamins.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Midazolam area under the plasma concentration-time curve from time 0 to 24 hours after dosing (AUC0-24) | Days 1-6
Midazolam maximum observed plasma concentration (Cmax) | Days 1-6
Omeprazole area under the plasma concentration-time curve from time 0 to 24 hours after dosing (AUC0-24) | Days 1-6
Omeprazole maximum observed plasma concentration (Cmax) | Days 1-6

SECONDARY OUTCOMES:
Telaprevir area under the plasma concentration-time curve from time 0 to 24 hours after dosing (AUC0-24) | Days 1-12
Telaprevir maximum observed plasma concentration (Cmax) | Days 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rice, MD, Principal Investigator — Spaulding Clinical
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States